CLINICAL TRIAL: NCT01225367
Title: Detection and Characterization of Cardio-pulmonary Patho-physiological States and Diseases by Ultrasound Transthoracic Doppler
Brief Title: The Use of a Ultra-sound of the Lung to Diagnose Lung Diseases
Status: Completed | Type: Observational
Sponsor: Echosense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ES_DOP05
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2011-05

CONDITIONS: Pulmonary Pathologies; Cardio-pulmonary Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulmonary doppler
  Interventions: Device: ultrasound doppler monitoring

INTERVENTIONS:
Device: ultrasound doppler monitoring — Regular noninvasive chest echo monitoring

SUMMARY:
The study is a prospective open evaluating study of Ultrasound/Doppler application to the chest cavity intended to detect and characterize pathologies of the pulmonary and cardio-vascular system.

The system is a noninvasive non-imaging device designated to monitor flow and movement velocity and display the data continuously.

ELIGIBILITY:
Inclusion Criteria:

* Age 18y or older
* patients who are clinically suspected of having a significant pulmonary or cardio-pulmonary disease
* Patients with CHF
* Patients with pulmonary hypertension
* Patients with COPD
* Patients with Asthma
* Signed informed consent
* Normal subjects

Exclusion Criteria:

* Patients with unstable conditions: unstable angina, uncontrolled CHF, etc
* Inability to assume a sitting or supine position
* Patients with severe chest wall deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Diagnose specific pattern of LDS signals as Power and Velocity in pulmonary diseases in comparison to controls. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Person, MD, Principal Investigator — Elisha Hospital
Locations (1):
- Elisha hospital, Haifa, Israel